CLINICAL TRIAL: NCT05319639
Title: Phase I/II Study of the Combination of Irinotecan and POF (Paclitaxel Plus Oxaliplatin Plus 5-fluorouracil Plus Leucovorin) and Tislelizumab
Brief Title: Phase I/II Study of the Combination of Irinotecan and POF (POFI) and Tislelizumab
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYLT-023
Record Dates: First submitted 2022-04-01; First posted 2022-04-08 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-01

CONDITIONS: Gastric Cancer Stage IV
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; Levoleucovorin; Fluorouracil; Paclitaxel; Irinotecan; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- POFI and Tislelizumab (Experimental): This study will include a sequential evaluation of 3 subjects per cohort. Irinotecan 135 → 150 and paclitaxel 45 → 67.5 → 90 mg/m2 on day 1.
  The rest of regimen is that oxaliplatin (85 mg/m2) and Lev-leucovolin (200 mg/m2).Subsequently, a 46-hour infusion of fluorouracil (2400 mg/m2) was administered using an ambulatory pump, repeating the cycle every 14 days. Tislelizumab 200mg，repeating the cycle every 14 days.
  A dose limiting toxicity (DLT) event is defined as any of the following events in the first 4-week period:
  CTCAE Grade 4 event (except for neutropenia lasting for ≤ 5 days); Grade 3 non-hematologic toxicity (except for nausea and vomiting that could be improved with optimal supportive care, escalation of alkaline phosphatase) If a DLT is experienced in any cohort, the cohort will be expanded to 6 subjects. If 2 DLTs are experienced in any cohort, the dose escalation ceased. The MTD was defined as the dose having at most two out of six patients experience DLT.
  Interventions: Drug: Oxaliplatin; Drug: Levo-Leucovorin; Drug: 5-fluorouracil; Drug: Paclitaxel; Drug: Irinotecan; Drug: Tislelizumab

INTERVENTIONS:
Drug: Oxaliplatin — Oxaliplatin will be administered on day 1 of each cycle at 85mg/m2 once every 14 days.
Drug: Levo-Leucovorin — Levo-Leucovorin will be administered on day 1 of each cycle at 200 mg/m2 once every 14 days.
Drug: 5-fluorouracil — 5-fluorouracil will be administered at 2400 mg/m2 over 46-hour every 14 days.
Drug: Paclitaxel — Paclitaxel will be administered on day 1 of each cycle at 45mg/m2 at dose level 1; 67.5 mg/m2 at dose level 2 ; 90 mg/m2 at dose level 3; 112.5 mg/m2 at dose level 4 once every 14 days.
Drug: Irinotecan — Irinotecan will be administered on day 1 of each cycle at 135 mg/m2 at dose level 1; 150 mg/m2 at dose level 2 once every 14 days.
Drug: Tislelizumab — Tislelizumab will be administered on day 1 of each cycle at 200mg once every 14 days.

SUMMARY:
The purpose of the phase I/II study is to establish the safety of Combination of Irinotecan and paclitaxel with 5-FU, leucovorin, oxaliplatin and Tislelizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced unresectable, histologically confirmed adenocarcinoma of the gastric or gastroesophageal junction.
2. With or without measurable lesions.
3. Patients must have a performance status of 0-1 on the Eastern Cooperative Oncology Group (ECOG) scale.
4. Without serious system dysfunction and could tolerate chemotherapy. With normal marrow, liver and renal function: a hemoglobin (HGB) of ≥100g/L (without blood transfusion during 14 days); a leucopenia count of ≥4.0×109/L; a platelet count of ≥100×109/L; a total bilirubin (TBil) of ≤1.5 upper normal limitation (UNL); a creatinine (Cr) of ≤ 1.5 UNL; a creatinine clearance rate ≥ 50ml/min (Cockcroft-Gault); a alanine aminotransferase (ALAT) and aspartate aminotransferase (ASAT) of ≤2.5 UNL or ≤5 UNL in case of liver metastasis.
5. Life expectancy ≥3 months.
6. With normal electrocardiogram results and no history of congestive heart failure.
7. With normal coagulation function: activated partial thromboplastin time (APTT), prothrombin time (PT) and INR, each ≤ 1.5 x ULN.
8. Female subjects of child-bearing potential must agree to use contraceptive measures starting 1 week before the administration of the first dose of Tislelizumab until 8 weeks after discontinuing study drug. Male subjects must agree to use contraceptive measures during the study and 8 weeks after last dose of study drug
9. With written informed consent signed voluntarily by patients themselves or their supervisors witted by doctors.
10. With good compliance and agree to accept follow-up of disease progression and adverse events.

Exclusion Criteria:

1. Patients with a history of another neoplastic disease within the past three years, excluding basal cell carcinoma of the skin, cervical carcinoma in situ, or nonmetastatic prostate cancer.
2. Patients with brain or central nervous system metastases, including leptomeningeal disease.
3. Pregnant (positive pregnancy test) or breast feeding.
4. Serious, non-healing wound, ulcer, or bone fracture.
5. Significant cardiac disease as defined as: unstable angina, New York Heart Association (NYHA) grade II or greater, congestive heart failure, history of myocardial infarction within 6 months Evidence of bleeding diathesis or coagulopathy.
6. History of a stroke or CVA within 6 months.
7. Clinically significant peripheral vascular disease.
8. Inability to comply with study and/or follow-up procedures.
9. Patients with any other medical condition or reason, in that investigator's opinion, makes the patient unstable to participate in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2023-02-16 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The maximum dose tolerated | 1 month
  To determine the maximum tolerated dose of POFI with different doses of irinotecan and paclitaxel combined with Tislelizumab in the first month.

SECONDARY OUTCOMES:
Overall Response Rate | 2 years
  Clinical response of treatment according to RESIST v1.1 criteria (ORR, objective response rate).
Progression-free survival | 2 years
  The length of time from enrollment until the time of progression of disease (PFS, progression-free survival).
Overall survival | 2 years
  The length of time from enrollment until the time of death (OS, overall survival).

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian cancer hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No